CLINICAL TRIAL: NCT06720935
Title: Contemporary Use of Coils During Percutaneous Coronary Intervention: From the Multicenter COILSEAL Registry
Brief Title: Use of Coils During Percutaneous Coronary Intervention
Acronym: COILSEAL
Status: Completed | Type: Observational
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Enrico Cerrato, Interventional Cardiologist, San Luigi Gonzaga Hospital
Other Study IDs: 002-2024
Record Dates: First submitted 2024-09-29; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Percutaneous Coronary Intervention (PCI); Coronary Artery Disease
Keywords: Coils; Coronary Artery Perforation; Coronary Fistulas; Coronary aneurysm
MeSH Terms: conditions — Coronary Artery Disease; Coronary Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing to percutaneous coronary intervention with coils: The study involves patients undergoing coils embolization for treating coronary artery perforation or coronary fistulas/aneurysm during percutaneous coronary intervention

SUMMARY:
Use of coils during percutaneous coronary interventions (PCI) is sometimes life-saving and useful althought currently off-label and with unknown clinical outcomes. The study aims to report and compare in-hospital and long-term outcomes of patients undergoing coils implantation for treating coronary perforation or closing coronary aneurysms/fistulas.

DETAILED DESCRIPTION:
Background. Use of coils during percutaneous coronary interventions (PCI) is sometimes life-saving and useful althought currently off-label and with unknown clinical outcomes Objectives. To report and compare in-hospital and long-term outcomes of patients undergoing coils implantation for treating coronary perforation or closing coronary aneurysms/fistulas.

Methods. Among 245.652 PCIs performed in 17 high-volume European centers, patients treated with coils will be identified.

The primary outcome was technical success, defined as the successful sealing coronary perforation or aneurysm/fistulas and procedural success defined as technical success without in-hospital Major Cardiovascular Events (MACe). Long-term MACE and mortality were also reported

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery perforation or coronary artery fistula/aneurysm suitable treating with coils embolization

Exclusion Criteria:

* Patients without coronary artery disease suitable of coils treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with coronary artery perforation or coronary fistula/aneurysm treated with coils embolization during percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
Rate of Technical Success | intraprocedural
  Rate of technical success is defined as effective sealing of coronary perforation or coronary fistulas/aneurysm after coils embolization

SECONDARY OUTCOMES:
Rate of Procedural success | Intraprocedural
  Rate of technical success without In Hospital Major Cardiovascular Events including death, target vessel myocardial infarction and re-PCI or CABG

CONTACTS AND LOCATIONS:
Locations (1):
- San Luigi Gonzaga Hospital, Orbassano, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided